CLINICAL TRIAL: NCT01436318
Title: Respiratory Muscle Strength and Function in Healthy Children
Brief Title: Respiratory Muscle Strength and Function in Healthy Kids
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: HK 176-2011
Record Dates: First submitted 2011-09-16; First posted 2011-09-19 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Respiratory Muscle Strength
Keywords: Healthy Kids; Respiratory; Volunteers

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Respiratory Function: Children will undergo one session of pulmonary function and strength testing

SUMMARY:
Respiratory muscle strength training (RMST) is a potential treatment option that has been shown to increase strength and ventilatory function in critically ill patients, patients on ventilators and patients with mild neuromuscular weakness. Currently researchers are examining the role of inspiratory muscle strength training (IMST) in pressure performance of ventilator dependent children with Pompe disease. However, normal pressure-flow-timing responses of lung function are not well-characterized in healthy children. The purpose of this study is to measure RMST-induced changes in respiratory function in healthy children. Children will undergo one session of lung function and strength testing. By studying healthy children's respiratory function, this study will also help to develop more efficient respiratory muscle training exercise prescriptions for children with neuromuscular weakness and impaired respiratory function.

DETAILED DESCRIPTION:
The goals of this study are to collect and evaluate respiratory muscle strength training (RMST) induced changes in ventilatory function in healthy children. Children will undergo one session of pulmonary function and strength testing to quantify rate of inspiratory and expiratory pressure development and to determine whether inspiratory and expiratory pressure correlate to maximal respiratory pressures and forced pulmonary function tests. Currently normal pressure-flow-timing responses are not well-characterized in healthy children. The purpose of this study is to help develop more efficient RMST exercise prescriptions for ill children on ventilators and with neuromuscular weakness.

Participants in the study will refrain from caffeine products and exercise on the day of respiratory testing. In conjunction with respiratory testing, baseline and exertional blood pressure, heart and respiratory rate, and pulse oximetry will be monitored. Participants will complete tidal flow-volume assessments and forced expiratory maneuvers according to the AMerican Thoracic Society guidelines. Participants will undergo 5 sets of 10 maximal-effort breaths against standardized resistances (one set each at 0, 5, 10, 15, and 20 cm H20). Following each set, subjects will rate the load magnitude and their feelings of breathing discomfort using a 0-10 visual analog scale. Participants will also perform maximal inspiratory and expiratory pressure maneuvers. All tests will be separated by at least 2-3 minutes of rest.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 4-16 years of age.
* Healthy subjects

Exclusion Criteria:

* Have primary pulmonary disease
* Have primary neuromuscular disease
* Have a connective tissue or autoimmune disease
* Have had a respiratory infection with in 15 days prior to study date
* Have acute aminoglycosides antibiotic therapy with in 15 days prior to study date
* Have acute corticosteroids with in 15 days prior to study date
* Have a need to use an inhaler routinely
* Have hepatic failure
* Have hematologic failure
* Have participated in other studies related to medications or exercise
* Have used tobacco products
* Have other precautions

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Children
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-04; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Testing | Day 1
  Subjects will complete tidal flow-volume assessments and forced expiratory maneuvers.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K Smith, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Ramonatxo M, Amsalem FA, Mercier JG, Jean R, Prefaut CG. Ventilatory control during exercise in children with mild or moderate asthma. Med Sci Sports Exerc. 1989 Feb;21(1):11-7. doi: 10.1249/00005768-198902000-00003. PMID 2494415
- [Background] Villafranca C, Borzone G, Leiva A, Lisboa C. Effect of inspiratory muscle training with an intermediate load on inspiratory power output in COPD. Eur Respir J. 1998 Jan;11(1):28-33. doi: 10.1183/09031936.98.11010028. PMID 9543266
- [Background] Tzelepis GE, Vega DL, Cohen ME, Fulambarker AM, Patel KK, McCool FD. Pressure-flow specificity of inspiratory muscle training. J Appl Physiol (1985). 1994 Aug;77(2):795-801. doi: 10.1152/jappl.1994.77.2.795. PMID 8002530
- [Background] Tzelepis GE, Kasas V, McCool FD. Inspiratory muscle adaptations following pressure or flow training in humans. Eur J Appl Physiol Occup Physiol. 1999 May;79(6):467-71. doi: 10.1007/s004210050538. PMID 10344453
- [Background] Coast JR, Jensen RA, Cassidy SS, Ramanathan M, Johnson RL Jr. Cardiac output and O2 consumption during inspiratory threshold loaded breathing. J Appl Physiol (1985). 1988 Apr;64(4):1624-8. doi: 10.1152/jappl.1988.64.4.1624. PMID 3378996
- [Background] Romer LM, McConnell AK. Specificity and reversibility of inspiratory muscle training. Med Sci Sports Exerc. 2003 Feb;35(2):237-44. doi: 10.1249/01.MSS.0000048642.58419.1E. PMID 12569211
- [Background] Otis AB. Pressure-flow relationships and power output of breathing. Respir Physiol. 1977 Jun;30(1-2):7-14. doi: 10.1016/0034-5687(77)90017-2. PMID 877452
- [Background] Mognoni P, Saibene F, Sant'Ambrogio G, Agostoni E. Dynamics of the maximal contraction of the respiratory muscles. Respir Physiol. 1968 Mar;4(2):193-202. doi: 10.1016/0034-5687(68)90051-0. No abstract available. PMID 5689337
- [Background] Read DJ, Freedman S, Kafer ER. Pressures developed by loaded inspiratory muscles in conscious and anesthetized man. J Appl Physiol. 1974 Aug;37(2):207-18. doi: 10.1152/jappl.1974.37.2.207. No abstract available. PMID 4853759
- [Background] Pengelly LD, Alderson AM, Milic-Emili J. Mechanics of the diaphragm. J Appl Physiol. 1971 Jun;30(6):797-805. doi: 10.1152/jappl.1971.30.6.797. No abstract available. PMID 5580797
- [Background] Ameredes BT, Zhan WZ, Prakash YS, Vandenboom R, Sieck GC. Power fatigue of the rat diaphragm muscle. J Appl Physiol (1985). 2000 Dec;89(6):2215-9. doi: 10.1152/jappl.2000.89.6.2215. PMID 11090570
- [Background] Goldman MD, Grassino A, Mead J, Sears TA. Mechanics of the human diaphragm during voluntary contraction: dynamics. J Appl Physiol Respir Environ Exerc Physiol. 1978 Jun;44(6):840-8. doi: 10.1152/jappl.1978.44.6.840. PMID 670007
- [Background] Fitting JW, Easton PA, Grassino AE. Velocity of shortening of inspiratory muscles and inspiratory flow. J Appl Physiol (1985). 1986 Feb;60(2):670-7. doi: 10.1152/jappl.1986.60.2.670. PMID 3081483
- [Background] Komarow HD, Myles IA, Uzzaman A, Metcalfe DD. Impulse oscillometry in the evaluation of diseases of the airways in children. Ann Allergy Asthma Immunol. 2011 Mar;106(3):191-9. doi: 10.1016/j.anai.2010.11.011. Epub 2011 Jan 6. PMID 21354020
- [Background] Younes M, Riddle W. A model for the relation between respiratory neural and mechanical outputs. I. Theory. J Appl Physiol Respir Environ Exerc Physiol. 1981 Oct;51(4):963-78. doi: 10.1152/jappl.1981.51.4.963. PMID 7298440
- [Background] Parthasarathy S, Jubran A, Laghi F, Tobin MJ. Sternomastoid, rib cage, and expiratory muscle activity during weaning failure. J Appl Physiol (1985). 2007 Jul;103(1):140-7. doi: 10.1152/japplphysiol.00904.2006. Epub 2007 Mar 29. PMID 17395760
- [Background] Butler JE. Drive to the human respiratory muscles. Respir Physiol Neurobiol. 2007 Nov 15;159(2):115-26. doi: 10.1016/j.resp.2007.06.006. Epub 2007 Jun 17. PMID 17660051
- [Background] Rowley KL, Mantilla CB, Sieck GC. Respiratory muscle plasticity. Respir Physiol Neurobiol. 2005 Jul 28;147(2-3):235-51. doi: 10.1016/j.resp.2005.03.003. PMID 15871925
- [Background] Osborne S, Road JD. Diaphragm and phrenic nerve activities during inspiratory loading in anesthetized rabbits. Respir Physiol. 1995 Mar;99(3):321-30. doi: 10.1016/0034-5687(94)00109-d. PMID 7770667
- [Background] American Thoracic Society; European Respiratory Society. ATS/ERS statement: raised volume forced expirations in infants: guidelines for current practice. Am J Respir Crit Care Med. 2005 Dec 1;172(11):1463-71. doi: 10.1164/rccm.200408-1141ST. No abstract available. PMID 16301301
- [Background] Polkey MI, Hamnegard CH, Hughes PD, Rafferty GF, Green M, Moxham J. Influence of acute lung volume change on contractile properties of human diaphragm. J Appl Physiol (1985). 1998 Oct;85(4):1322-8. doi: 10.1152/jappl.1998.85.4.1322. PMID 9760323